CLINICAL TRIAL: NCT06303375
Title: Effect of Kinesio Taping on Pain, Posture and Function in Patient With Lower Cross Syndrome
Brief Title: Effect of Kinesio Taping on Pain, Posture and Function in Lower Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01718 Nida Kausar
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lower Cross Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping along with conventional physical therapy (Experimental): treatment with moist hot pack along with stretching of tight erector spinae, hip flexors and strengthening of weak abdominals and gluteal muscles along with Kinesiotaping using inhibition and facilitation technique for LCS.
  Interventions: Other: Kinesio taping; Other: Conventional physical therapy
- conventional physical therapy (Active Comparator): Treatment with moist hot pack along with stretching of tight erector spinae, hip flexors and strengthening of weak abdominals and gluteal muscles.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Kinesio taping — Kinesiotaping using inhibition technique in tight muscles and facilitation technique in weak muscles for LCS. Treatment sessions 3 days per week for almost 04 weeks.
  10 mins moist hot pack
  * Stretching exercises of tight erector spinae, hip flexors 3-4 times a week 5 sec hold 5-7 reps 1 set.
  * Strengthening of weak abdominals and gluteal muscles 2-3 times in a week
  Arms: Kinesio taping along with conventional physical therapy
Other: Conventional physical therapy — 10 mins moist hot pack
  * Stretching exercises of tight erector spinae, hip flexors 3-4 times a week 5 sec hold 5-7 reps 1 set.
  * Strengthening of weak abdominals and gluteal muscles 2-3 times in a week

SUMMARY:
Determine the impact of Kinesio taping on pain, postural alignment and functional outcomes in individuals with lower cross syndrome.

DETAILED DESCRIPTION:
Participants with lower cross syndrome who present to physical therapy department will be screened for eligibility on basis of inclusion and exclusion criteria. Group A will receive the treatment with moist hot pack along with stretching of tight erector spinae, hip flexors and strengthening of weak abdominals and gluteal muscles along with Kinesiotaping using inhibition and facilitation technique for LCS and Group B will receive the treatment with moist hot pack along with stretching of tight erector spinae, hip flexors and strengthening of weak abdominals and gluteal muscles. The patients will receive the treatment sessions 3 days per week for almost 04 weeks. They will be evaluated after the treatment for PAIN, POSTURAL ASSESSMENT, FUNCTIONAL DISABILITY in order to check for the effect of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age- 30 to 50 years.
* Female patients.
* Anterior pelvic tilting > 7-10 degrees.
* Postural imbalance characterized by anterior pelvic tilt, lumbar hyper lordosis, and associated muscle imbalances.
* Discomfort, pain, or limitations related to the lower back, pelvis, and hips attributed to LCS.
* Willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Musculoskeletal pathologies affecting the lower back, pelvis, hips, or lower extremities (e.g., herniated disc, lumbar radiculopathy, lumbar stenosis, hip labral tear).
* Kinesiotaping interventions for LCS in the past 3 months.
* Allergies to tape materials or skin sensitivities that might prevent safe tape application.
* Pregnant individuals due to potential discomfort.
* Open wounds, infections, or skin conditions at the taping application site.
* Severe cardiovascular, pulmonary, renal, or neurological diseases.
* In other clinical trials involving interventions for LCS.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 4th week
  To assess pain using a Visual Analog Scale (VAS), provide patient with a straight line ranging from "No Pain "to "Worst pain Imaginable "Ask patient to mark a point on line that represents their current pain intensity, with understanding that the left end means no pain, and the right end means the most severe pain imaginable, measure distance in millimeters from "No pain "end to the marked point to quantify the pain level. Pain is assess at the end of every week.
Anterior pelvic tilting | 4th week
  The hand-held pelvic inclinometer's is use for measure anterior pelvic tilting. Anterior pelvic tilting is measure at the end of every week.
Oswestry Disability Index (ODI) | 4th week
  The Oswestry Disability Index (ODI) is a widely used questionnaire to assess the functional disability and impact of lower back pain on an individual's daily life. Patients are asked to rate their level of disability on a scale from 0 to 5, with 0 indicating no disability and 5 indicating the highest level of disability. It is divided into ten sections that each target various tasks or functions. Higher percentages indicate greater disability. Functional disability through ODI assess after every 2nd week.
Muscle Length | 4th week
  The length of the bilateral Iliopsoas muscle was measured using a Universal Goniometer and the Modified Thomas test. A non-elastic measuring tape was used to examine the length of the spinal extensor muscle. Abdominal muscular strength and bilateral Gluteus maximus Manual muscle testing was graded according to the MRC grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No